CLINICAL TRIAL: NCT01000805
Title: A Phase 4, 8-Week, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Efficacy of Duloxetine 60 mg Once Daily in Outpatients With Major Depressive Disorder and Associated Painful Physical Symptoms
Brief Title: A Study of Duloxetine in Major Depressive Disorder (MDD) and Associated Painful Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13399; F1J-US-HMGR (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2011-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Participants received 30 mg duloxetine once daily (QD) by mouth (po) for 1 week followed by 60 mg QD, po for 7 weeks.
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine
Drug: Placebo — Participants received placebo QD, po for 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if 60 mg of duloxetine given once a day by mouth for 8 weeks to patients diagnosed with major depressive disorder, who also report associated painful physical symptoms, is better than placebo when treating depression and its associated painful symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Major Depressive Disorder (MDD) as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and confirmed by Mini International Neuropsychiatric Interview (MINI)
* Montgomery-Asberg Depression Rating Scale (MADRS) total score of greater than or equal to 20 during the Screening Phase
* At least 1 previous episode of depression
* Painful physical symptoms with a score greater than or equal to 3 on the Brief Pain Inventory-Short Form (BPI-SF) average pain question during the Screening Phase
* A Clinical Global Impression of Severity (CGI-S) score of greater than or equal to 4 during the Screening Phase
* Written informed consent

Exclusion Criteria:

* Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device
* Previously completed or withdrawn from this study or any other study investigating duloxetine
* Women of child-bearing potential who are not using a medically accepted means of contraception
* Any current (within the past 6 months) DSM-IV-TR primary Axis I diagnosis other than MDD
* History of alcohol abuse or dependence within 1 year immediately prior to being screened for the study
* Any prior history of bipolar disorder, psychosis, or schizophrenia
* Have an Axis II disorder that would interfere with study compliance
* Lack of a response of any (lifetime of subject) episode of major depression greater than or equal to 2 adequate courses of antidepressant therapy, defined as a clinically appropriate dose for a minimum of 4 weeks or, alternatively, in the judgment of the investigator, the subject meets criteria for treatment-resistant depression
* Have previously received treatment of MDD or Generalized Anxiety Disorder (GAD) with an adequate trial of duloxetine and did not respond or could not tolerate duloxetine
* Diagnosis of acute liver injury or severe cirrhosis
* Uncontrolled narrow-angle glaucoma
* Positive urine drug screen for any substance of abuse.
* A serious medical illness, including any cardiovascular, hepatic, renal, respiratory, hematologic, endocrinologic, or neurologic disease, or a clinically significant laboratory abnormality that is not stabilized or is anticipated to require intervention
* A history of substance abuse or dependence within 1 year before being screened for the study
* History of a serious suicide attempt or subject judged clinically to be at serious suicidal risk
* Require continuous use of opioid analgesics for 6 or more months because of chronic pain
* Pain of a known origin
* Meets criteria for fibromyalgia as defined by the American College of Rheumatology
* Experiences greater than or equal to 1 migraine headache per week
* Have had electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), or vagus nerve stimulation (VNS) within 1 year prior to being screened for the study
* Initiating, changing, or stopping psychotherapy within 6 weeks prior to being screened for the study or at any time during the study
* Investigator or subject anticipates initiating, changing, or stopping non-pharmacologic or alternative therapies for painful physical symptoms at any time during the study
* Are taking any excluded medications within 7 days prior to randomization with the exception of fluoxetine which cannot be taken within 30 days prior to randomization
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to randomization or have the potential need to use an MAOI during the study or within 5 days of discontinuing study drug
* Frequent and/or severe allergic reactions with multiple medications
* Abnormal thyroid stimulating hormone concentration
* Has epilepsy or history of seizure disorder or received treatment with anticonvulsant medication for epilepsy or seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brown Deer, Wisconsin
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arcachon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Élancourt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulon
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzenau in Unterfranken
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ellwangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgovişte
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Luleå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm

REFERENCES:
- [Background] Dmitrienko A, Offen WW, Westfall PH. Gatekeeping strategies for clinical trials that do not require all primary effects to be significant. Stat Med. 2003 Aug 15;22(15):2387-400. doi: 10.1002/sim.1526. PMID 12872297
- [Derived] Gaynor PJ, Gopal M, Zheng W, Martinez JM, Robinson MJ, Marangell LB. A randomized placebo-controlled trial of duloxetine in patients with major depressive disorder and associated painful physical symptoms. Curr Med Res Opin. 2011 Oct;27(10):1849-58. doi: 10.1185/03007995.2011.609539. Epub 2011 Aug 12. PMID 21838411

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 262 | 266
Completed | 192 | 204
Not Completed | 70 | 62
Not completed — Adverse Event | 21 | 9
Not completed — Lack of Efficacy | 5 | 16
Not completed — Lost to Follow-up | 16 | 21
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 12 | 8
Not completed — Withdrawal by Subject | 16 | 6
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 262 | 266 | 528
Age Continuous [Mean (Standard Deviation); unit: years] | 46.15 (13.27) | 45.73 (12.85) | 45.94 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 184 | 364
  Male | 82 | 82 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 63 | 131
  Not Hispanic or Latino | 194 | 203 | 397
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 47 | 78
  White | 222 | 213 | 435
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 18 | 16 | 34
  France | 29 | 33 | 62
  Puerto Rico | 37 | 35 | 72
  Romania | 11 | 15 | 26
  Sweden | 22 | 22 | 44
  United States | 145 | 145 | 290
Brief Pain Inventory Severity: Worst Pain Score (BPI-S: Worst Pain) [Mean (Standard Deviation); unit: units on a scale] — The BPI-S: Worst Pain is a self-reported scale that measures the severity of pain based on the worst pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 6.93 (1.65) | 6.86 (1.70) | 6.89 (1.67)
Brief Pain Inventory Severity: Least Pain Score (BPI-S: Least Pain) [Mean (Standard Deviation); unit: units on a scale] — The BPI-S: Least Pain is a self-reported scale that measures the severity of pain based on the least pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 4.27 (2.17) | 4.11 (2.22) | 4.19 (2.19)
Brief Pain Inventory Severity: Average Pain Score (BPI-S: Average Pain) [Mean (Standard Deviation); unit: units on a scale] — The BPI-S: Average Pain is a self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 5.68 (1.69) | 5.58 (1.67) | 5.63 (1.68)
Brief Pain Inventory Severity: Pain Right Now Score (BPI-S: Pain Right Now) [Mean (Standard Deviation); unit: units on a scale] — The BPI-S: Pain Right Now is a self-reported scale that measures the severity of pain based on the pain right now. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 5.29 (2.37) | 5.34 (2.10) | 5.32 (2.24)
Brief Pain Inventory - Interference (BPI-I) [Mean (Standard Deviation); unit: units on a scale] — The BPI-I scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
  units on a scale | 5.65 (2.20) | 5.67 (2.11) | 5.66 (2.16)
Clinical Global Impressions of Severity Scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — The CGI-S measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 4.58 (0.63) | 4.58 (0.63) | 4.58 (0.63)
Montgomery Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
  units on a scale | 29.91 (4.92) | 30.39 (5.25) | 30.15 (5.09)
Sheehan Disability Scale-Item 1 (SDS-Item 1), N=196,200,396 [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and Item 1 is used to assess the effect of the participant's symptoms on their work/school schedule. Scores range from 0 to 10 with higher values indicating greater disruption in the participant's work/school life.
  units on a scale | 6.24 (2.30) | 6.23 (2.15) | 6.23 (2.22)
Sheehan Disability Scale-Item 2 (SDS-Item 2), N=262,265,527 [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and Item 2 is used to assess the effect of the participant's symptoms on their social life/leisure activities. Scores range from 0 to 10 with higher values indicating greater disruption in the patient's social life.
  units on a scale | 6.43 (2.27) | 6.50 (2.15) | 6.46 (2.21)
Sheehan Disability Scale-Item 3 (SDS-Item 3), N=262,265,527 [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and Item 3 is used to assess the effect of the participant's symptoms on their family life/home responsibilities. Scores range from 0 to 10 with higher values indicating greater disruption in the participant's family life/home responsibilities.
  units on a scale | 6.42 (2.21) | 6.45 (2.06) | 6.44 (2.13)
Sheehan Disability Scale -Total Score (SDS Total), N=262,265,527 [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life.
  units on a scale | 19.16 (6.00) | 19.38 (5.84) | 19.27 (5.92)
Number of Previous Major Depressive Disorder (MDD) Episodes [Mean (Standard Deviation); unit: number of previous episodes] | 3.52 (3.98) | 3.67 (4.88) | 3.60 (4.45)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Brief Pain Inventory-Short Form (BPI-SF) Average Pain Score During the 8-week Treatment Period
Description: A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). The overall change is based on the estimated main treatment effect. The Least Squares (LS) Mean Value was adjusted for treatment, investigator, visit, baseline, treatment*visit interaction, and baseline*visit interaction.
Time Frame: Day 1 through 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 261
units on a scale | -1.93 (0.11) | -1.31 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This p-value is for the main effect of treatment; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.90 to -0.33]

2. Primary Outcome: Change From Baseline in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score at Week 8
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). The Least Squares (LS) Mean Value was adjusted for treatment, investigator, visit, baseline, treatment*visit interaction, and baseline*visit interaction.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine: Participants received 30 mg duloxetine once daily (QD) by mouth (po) for 1 week, followed by 60 mg QD, po for 7 weeks.
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 262
units on a scale | -16.77 (0.67) | -12.73 (0.64)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.04, 95% CI 2-sided [-5.83 to -2.24]

3. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Total and Item Scores at Week 8
Description: SDS is completed by participant; used to assess effect of the participant's symptoms on their work/social/family life. Total scores range from 0 to 30; higher values indicate greater disruption in the participant's work/social/family life. Each item score ranges from 0 to 10 with higher values indicating greater disruption in the participant's work/school life (item 1), social life/leisure activities (item 2), or family life/home responsibilities (item 3). The LS Mean Value was adjusted for treatment, investigator, visit, baseline, treatment*visit interaction, and baseline*visit interaction.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 250 | 260
units on a scale
  Disrupt Work/School Work (N=182, 196) | -2.82 (0.22) | -2.36 (0.20)
  Disrupt Social Life/Leisure Activities | -3.04 (0.19) | -2.31 (0.18)
  Disrupt Family/Home Responsibilities | -3.02 (0.19) | -2.49 (0.18)
  SDS Total Score | -8.88 (0.54) | -7.13 (0.52)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.112, Mixed Models Analysis — This is the p-value for the Disrupt Work/School Work score; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.03 to 0.11]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — This the p-value for the Disrupt Social Life/Leisure score; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.24 to -0.22]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis — This is the p-value for the Disrupt Family Life/Home score; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.04 to -0.02]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis — P-value for the SDS Total score. First gated secondary outcome measure. Gatekeeper strategy controlled experiment-wise type I error for 5 secondary outcomes with stepwise comparisons of treatments until outcome failed to be significant (p>0.05); Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-3.20 to -0.29]

4. Secondary Outcome: Change From Baseline in the Percentage of Participants Achieving Remission up to Week 8
Description: The Montgomery Asberg Depression Rating Scale (MADRS) is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Remission is defined as achieving a MADRS total score ≤12.
Time Frame: Baseline, up to 8 weeks
Population: All randomized participants with a post-baseline result, Last Observation Carried Forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 262
percentage of participants | 47.0 | 32.8
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — This is the second gated secondary outcome measure. A gatekeeper strategy (Dmitrienko et al. 2003) controlled experiment-wise type I error for 5 secondary outcomes. Treatments were compared stepwise until an outcome failed to be significant (p>0.05)

5. Secondary Outcome: Percentage of Participants Achieving Remission up to Week 8
Description: The Montgomery Asberg Depression Rating Scale (MADRS) is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale from 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Remission is defined as achieving a MADRS total score ≤12 at the last 2 nonmissing consecutive visits (for example, visit 3 [week 1] and visit 4 [week 2], or visit 4 [week 2] and visit 5 [week 4], or visit 5 [week 4] and visit 6 [week 8]).
Time Frame: Up to 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 262
percentage of participants | 29.5 | 18.7
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0082, Cochran-Mantel-Haenszel — This is the third gated secondary outcome measure. A gatekeeper strategy (Dmitrienko et al. 2003) controlled experiment-wise type I error for 5 secondary outcomes. Treatments were compared stepwise until an outcome failed to be significant (p>0.05)

6. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at Week 4
Description: The MADRS is a rating scale for severity of depressive mood and symptoms. The MADRS has a 10-item checklist. Items are rated on a scale from 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). The Least Squares (LS) Mean Value was adjusted for treatment, investigator, visit, baseline, treatment*visit interaction, and baseline*visit interaction.
Time Frame: Baseline, 4 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 262
units on a scale | -14.15 (0.58) | -10.49 (0.55)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the fourth gated secondary outcome measure. A gatekeeper strategy (Dmitrienko et al. 2003) controlled experiment-wise type I error for 5 secondary outcomes. Treatments were compared stepwise until an outcome failed to be significant (p>0.05); Mean Difference (Final Values) = -3.66, 95% CI 2-sided [-5.20 to -2.11]

7. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at Week 2
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range from 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). The Least Squares (LS) Mean Value was adjusted for treatment, investigator, visit, baseline, treatment*visit interaction, and baseline*visit interaction.
Time Frame: Baseline, 2 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 262
units on a scale | -9.90 (0.49) | -7.71 (0.47)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — This is the fifth gated secondary outcome measure. A gatekeeper strategy (Dmitrienko et al. 2003) controlled experiment-wise type I error for 5 secondary outcomes. Treatments were compared stepwise until an outcome failed to be significant (p>0.05); Mean Difference (Final Values) = -2.19, 95% CI 2-sided [-3.50 to -0.89]

8. Secondary Outcome: Change From Baseline in the Brief Pain Inventory Severity and Interference Scores (BPI-S/BPI-I) at Week 8
Description: Measures pain severity and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference=average of nonmissing scores of individual interference items. LS Mean Value adjusted for treatment, investigator, visit, baseline, treatment*visit interaction, and baseline*visit interaction.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 261
units on a scale
  BPI Severity for Worst Pain | -2.25 (0.13) | -1.60 (0.12)
  BPI Severity for Least Pain | -1.48 (0.11) | -0.86 (0.10)
  BPI Severity for Average Pain | -1.93 (0.11) | -1.31 (0.10)
  BPI Severity for Pain Right Now | -2.00 (0.12) | -1.27 (0.12)
  BPI Pain Interference with General Activity | -2.01 (0.13) | -1.33 (0.13)
  BPI Pain Interference with Mood | -2.49 (0.14) | -1.76 (0.13)
  BPI Pain Interference with Walking Ability | -1.52 (0.13) | -1.06 (0.12)
  BPI Pain Interference with Normal Work | -2.02 (0.13) | -1.46 (0.13)
  BPI Pain Interference with Relations With Others | -2.01 (0.13) | -1.31 (0.13)
  BPI Pain Interference with Sleep | -1.94 (0.14) | -1.56 (0.14)
  BPI Pain Interference with Enjoyment of Life | -2.44 (0.14) | -1.77 (0.13)
  BPI Mean Pain Interference Score | -2.03 (0.12) | -1.46 (0.12)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Severity for Worst Pain score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-0.97 to -0.32]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for main effect of treatment for the BPI Severity for Least Pain score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.90 to -0.34]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Severity for Average Pain score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.90 to -0.33]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Severity for Pain Right Now score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.06 to -0.42]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Pain Interference with General Activity score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.03 to -0.33]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Pain Interference with Mood score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.09 to -0.37]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Pain Interference with Walking Ability score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.79 to -0.11]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Pain Interference with Normal Work score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.91 to -0.21]
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Pain Interference with Relations with Others score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.06 to -0.35]
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.042, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Pain Interference with Sleep score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.76 to -0.01]
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Pain Interference with Enjoyment of Life score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.03 to -0.31]
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the main effect of treatment for the BPI Mean Pain Interference score. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.88 to -0.25]

9. Secondary Outcome: Patient's Global Impressions of Improvement Scale (PGI-I) at Week 8
Description: A scale that measures the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). The Least Squares (LS) Mean Value was adjusted for treatment, investigator, visit, and treatment*visit interaction.
Time Frame: 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 195 | 211
units on a scale | 2.56 (0.08) | 3.04 (0.08)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.71 to -0.26]

10. Secondary Outcome: Number of Participants With Suicidal Behaviors, Ideations, and Acts Based on the Columbia Suicide Severity Rating Scale (C-SSRS) During the Double-blind Treatment Phase
Description: The C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of participants with suicidal behaviors, ideations, and acts are provided. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, and completed suicide. Suicidal ideation: a "yes" answer to any 1 of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation. Suicidal acts: a "yes" answer to actual attempt or completed suicide.
Time Frame: Baseline through 8 weeks
Population: All randomized participants with at least 1 post-baseline C-SSRS result.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 262
participants
  Suicidal Ideation | 26 | 41
  Suicidal Behavior | 1 | 0
  Suicidal Acts | 2 | 0
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.293, Fisher Exact — This is the p-value for suicidal ideation. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05

11. Other Pre Specified Outcome: Number of Participants With Abnormal Laboratory Values During the Double-blind Treatment Phase - High Alanine Amino Transferase/Serum Glutamate Pyruvate Transaminase (ALT/SGPT)
Description: Laboratory assessment of ALT/SGPT during the double-blind treatment phase. Normal ALT/SGPT ranges for males are 6.00 units per liter (U/L) (low) to 43.00 U/L (high). Normal ALT/SGPT ranges for females are 6.00 U/L (low) to 34.00 U/L (high).
Time Frame: Baseline through 8 weeks
Population: All randomized participants with a normal baseline (respective to the specified direction) and at least 1 post-baseline result.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 182 | 193
participants | 14 | 5
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.033, Fisher Exact — P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05

12. Secondary Outcome: Change From Baseline in Pulse Rate up to Week 8
Description: The change from baseline in pulse rate at week 8 is the primary analysis. For the primary analysis of pulse rate, the Least Squares (LS) Mean Value was adjusted for treatment, investigator, baseline, treatment*visit interaction, and baseline*visit interaction.
  The change from baseline in pulse rate up to week 8 is the secondary analysis. The LS Mean Value was adjusted for treatment, investigator, and baseline.
Time Frame: Baseline, up to week 8
Population: Primary analysis: All randomized participants with a baseline and at least 1 post-baseline result.
  Secondary analysis: Intention-to-treat population (ITT) with nonmissing baseline value and at least 1 nonmissing post-baseline value, LOCF.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 250 | 262
beats per minute (bpm)
  Change from Baseline in Pulse Rate at Week 8 | 1.58 (0.59) | -1.34 (0.57)
  Change from Baseline in Pulse Rate up to Week 8 | 1.71 (0.54) | -0.70 (0.53)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the Change from Baseline at Week 8. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 2.92, 95% CI 2-sided [1.34 to 4.51]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — This is the p-value for the Change up to Week 8. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 2.40, 95% CI 2-sided [0.97 to 3.83]

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Up to Week 8
Description: The change from baseline in SBP and DBP at week 8 is the primary analysis. For the primary analysis of SBP and DBP, the Least Squares (LS) Mean Value was adjusted for treatment, investigator, baseline, treatment*visit interaction, and baseline*visit interaction.
  The change from baseline in SBP and DBP up to week 8 is the secondary analysis. The LS Mean Value was adjusted for treatment, investigator, and baseline.
Time Frame: Baseline, up to week 8
Population: Primary analysis: All randomized participants with a baseline and at least 1 post-baseline result.
  Secondary analysis: Intention-to-treat population (ITT) with nonmissing baseline value and at least 1 nonmissing post-baseline value, Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 250 | 262
mm Hg
  Change from Baseline in SBP at Week 8 | 1.38 (0.80) | -0.52 (0.77)
  Change from Baseline in DBP at Week 8 | 0.52 (0.53) | 0.05 (0.51)
  Change from Baseline in SBP up to Week 8 | 1.41 (0.74) | -0.12 (0.72)
  Change from Baseline in DBP up to Week 8 | 0.31 (0.49) | 0.01 (0.48)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.083, Mixed Models Analysis — This is the p-value for the Change from Baseline in SBP at Week 8. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 1.90, 95% CI 2-sided [-0.25 to 4.04]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.513, Mixed Models Analysis — This is the p-value for the Change from Baseline in DBP at Week 8. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.95 to 1.90]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.124, ANCOVA — This is the p-value for the Change from Baseline in SBP up to Week 8. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 1.53, 95% CI 2-sided [-0.42 to 3.47]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.638, ANCOVA — This is the p-value for the Change from Baseline in DBP up to Week 8. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-0.98 to 1.60]

14. Secondary Outcome: Change From Baseline in Weight up to Week 8
Description: The change from baseline in weight at week 8 is the primary analysis. For the primary analysis of weight, the Least Squares (LS) Mean Value was adjusted for treatment, investigator, baseline, treatment*visit interaction, and baseline*visit interaction.
  The change from baseline in weight up to week 8 is the secondary analysis. The LS Mean Value was adjusted for treatment, investigator, and baseline.
Time Frame: Baseline, up to week 8
Population: Primary analysis: All randomized participants with a baseline and at least 1 post-baseline result.
  Secondary analysis: All randomized participants with a baseline and at least 1 nonmissing post-baseline result, Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 251 | 262
kilograms (kg)
  Change from Baseline in Weight at Week 8 | -0.77 (0.15) | 0.19 (0.15)
  Change from Baseline in Weight up to Week 8 | -0.74 (0.14) | 0.14 (0.13)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.37 to -0.54]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — This is the p-value for the Change from Baseline up to Week 8. P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.24 to -0.51]

ADVERSE EVENTS:
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 5/262 | 1/266
Other Adverse Events (participants affected / at risk) | 162/262 | 137/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=262) | Placebo (N=266)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=262) | Placebo (N=266)
Vision blurred (Eye disorders) | 7 (7) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 7 (8) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 6 (6)
Constipation (Gastrointestinal disorders) | 17 (18) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 15 (17) | 16 (16)
Dry mouth (Gastrointestinal disorders) | 22 (24) | 14 (14)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 2 (2)
Nausea (Gastrointestinal disorders) | 51 (55) | 24 (25)
Vomiting (Gastrointestinal disorders) | 7 (7) | 0 (0)
Fatigue (General disorders) | 11 (12) | 7 (7)
Irritability (General disorders) | 2 (2) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 13 (14) | 5 (5)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Dizziness (Nervous system disorders) | 13 (13) | 10 (10)
Headache (Nervous system disorders) | 30 (35) | 22 (28)
Somnolence (Nervous system disorders) | 24 (25) | 8 (8)
Anxiety (Psychiatric disorders) | 8 (8) | 5 (5)
Insomnia (Psychiatric disorders) | 11 (11) | 9 (9)
Yawning (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14 (15) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days